CLINICAL TRIAL: NCT01339767
Title: Markers of Autism Spectrum Disorders in At-Risk Toddlers: A Pilot Study
Brief Title: Study of Toddlers With Language Delay
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110144; 11-M-0144
Record Dates: First submitted 2011-04-20; First posted 2011-04-21 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2017-06-30

CONDITIONS: Autism; Language Acquisition; Language Development; Toddlers
Keywords: Autism; Language Acquisition; Language Development; Toddlers
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to learn more about risk factors for autism by studying the behavior and brain functioning of toddlers with early communication delays and typically developing toddlers. Children 12 or 18 months of age with language delays (i.e., no words at 18 months, limited vocalizations at 12 months) and typically developing toddlers may be eligible to participate. This study will be conducted at the NIH Clinical Center in Bethesda, Maryland. There will be an initial screening evaluation that will include behavioral assessment. Eligible participants will then complete a baseline visit that includes an overnight sleep study that includes Electroencephalogram (EEG) test to measure brain electrical activity, and an MRI scan. Follow-up visits that include behavioral assessment will occur every 6-12 months, depending on age at study entry. The final study visit will occur at 36 months of age and will include behavioral assessment, sleep/EEG study, and MRI. There is no cost for participation. Compensation will be provided. To find out if your child qualifies or for more information, please call 301-451-7822 (TTY: 1-866-411-1010) or e-mail NIMH-ASD@mail.nih.gov. National Institute of Mental Health, National Institutes of Health, Department of Health & Human Services.

DETAILED DESCRIPTION:
Objective

This investigation will focus on two areas: 1) early communication impairments as predictors of autism spectrum disorder (ASD) and later developmental delays, and 2) the relationship between communication and evidence of CNS function (sleep, EEG) and structure (MRI DTI and volumetrics) in young children at risk for ASD. The objective is to delineate early communicative impairments that predict ASD vs. other developmental delays and to examine how these impairments correlate with brain abnormalities in both structure and function.

Study Population

We will recruit 64 children [n=32 at 12 months of age (plus or minus 2 months); n=32 at 18 months of age (plus or minus 2 months)] who are at-risk for ASD due to communication/language delays (at-risk group). The at-risk children will be matched at initial on chronological age, SES, and sex, to typically developing children (n=75) with no history of developmental delays. These 139 participants will hereafter be referred to as the toddler sample. At the 36 month final visit, diagnostic status (e.g. ASD, non-ASD specific delays, catch up) will be determined for children in the at-risk group. In addition, 10 healthy adults, aged 18-40 will serve as control participants for the purpose of piloting the functional paradigms for the MRI portion of the protocol.

Design

We propose to conduct a prospective, longitudinal study of toddlers at-risk for ASD compared to typically developing toddlers. Children will complete behavioral testing and an overnight Sleep/EEG as well as MRI at either a 12 or 18 month initial. Follow-up visits that include behavioral assessment will occur at 24 and 36 months for all children (and at 18 months of age for the 12-month cohort). The Sleep/EEG and MRI will be repeated at the 36 month final follow-up.

Outcome Measures

Autism symptoms, language status, and cognitive development at 36 months will serve as the primary outcome measures.

ELIGIBILITY:
* INCLUSION CRITERIA:

At-risk Group:

1. 12 or 18 months of age (plus or minus 3 months)
2. Limited spoken words (for both the 12 and 18 month groups)
3. Expressive and Receptive scores in the Very Low range on the Mullen Scales of Early Learning (a standardized observational measure),

Typically Developing Group:

1. 12 or 18 months of age (plus or minor 3 months)
2. Development in nonverbal and verbal areas within age expectations (per scores on all 4 domains of the Mullen Scales of Early learning no more than 1.5 standard deviation below the mean).

Healthy Adult Group:

1. 18-40 years old

EXCLUSION CRITERIA:

At-risk Group:

1. Primary language spoken in the home is other than English
2. Prematurity at birth (defined as less than 36 weeks gestation), or birth weight significantly below normal for gestational age (SGA- small for gestational age) or other significant birth trauma.
3. Motor or other medical impairment deemed responsible for delays (e.g. cerebral palsy; known genetic disorder)

Typically Developing Group:

1. Primary language spoken in the home is other than English
2. Prematurity at birth (defined as less than 36 weeks gestation); or birth weight significantly below normal for gestational age (SGA- small for gestational age).
3. Motor or other medical impairment that would interfere with study participation
4. Known genetic disorder
5. Status as a younger sibling of a child diagnosed with autism

Healthy Adult Group:

1. Historical or current psychiatric, neurological, or serious medical illness
2. Primary language is other than English
3. Difficulty hearing (as some sounds and words will be presented during the MRI scan)
4. Head injury with loss of consciousness in the last year
5. Metal in the body which would make having an MRI scan unsafe, such as pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent eye liner or small metal fragments in the eye that welders and other metal workers may have.
6. Discomfort in small closed spaces (have claustrophobia) so that there would be discomfort in the MRI machine.
7. Inability to lie comfortably flat on the back for up to 60 minutes in the MRI scanner
8. If female, and pregnant
9. Inability to provide own consent

Ages: 9 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2011-04-18; Study Completion 2017-06-30

CONTACTS AND LOCATIONS:
Overall Officials: Audrey E Thurm, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Buschmann A, Jooss B, Rupp A, Dockter S, Blaschtikowitz H, Heggen I, Pietz J. Children with developmental language delay at 24 months of age: results of a diagnostic work-up. Dev Med Child Neurol. 2008 Mar;50(3):223-9. doi: 10.1111/j.1469-8749.2008.02034.x. Epub 2008 Feb 11. PMID 18266869
- [Background] Chawarska K, Klin A, Paul R, Volkmar F. Autism spectrum disorder in the second year: stability and change in syndrome expression. J Child Psychol Psychiatry. 2007 Feb;48(2):128-38. doi: 10.1111/j.1469-7610.2006.01685.x. PMID 17300551
- [Background] Dager SR, Wang L, Friedman SD, Shaw DW, Constantino JN, Artru AA, Dawson G, Csernansky JG. Shape mapping of the hippocampus in young children with autism spectrum disorder. AJNR Am J Neuroradiol. 2007 Apr;28(4):672-7. PMID 17416819
- [Derived] Hong X, Farmer C, Kozhemiako N, Holmes GL, Thompson L, Manwaring S, Thurm A, Buckley A. Differences in sleep EEG coherence and spindle metrics in toddlers with and without receptive/expressive language delay: a prospective observational study. J Neurodev Disord. 2025 Feb 22;17(1):11. doi: 10.1186/s11689-024-09586-1. PMID 39987026
- [Derived] Hong X, Farmer C, Kozhemiako N, Holmes GL, Thompson L, Manwaring S, Thurm A, Buckley A. Differences in Sleep EEG Coherence and Spindle Metrics in Toddlers With and Without Language Delay: A Prospective Observational Study. Res Sq [Preprint]. 2024 Feb 14:rs.3.rs-3904113. doi: 10.21203/rs.3.rs-3904113/v1. PMID 38410470
- [Derived] Smith EG, Condy E, Anderson A, Thurm A, Manwaring SS, Swineford L, Gandjbakhche A, Redcay E. Functional near-infrared spectroscopy in toddlers: Neural differentiation of communicative cues and relation to future language abilities. Dev Sci. 2020 Nov;23(6):e12948. doi: 10.1111/desc.12948. Epub 2020 Mar 20. PMID 32048419